CLINICAL TRIAL: NCT06040944
Title: The Effect of Antipsychotic Medication and the Associated Hyperprolactinemia as Risk Factor for Periodontal Diseases in Schizophrenic Patients: a Cohort Retrospective Study
Brief Title: Antipsychotic Induced Hyperprolactinemaia as Risk Factor for Periodontitis in Schizophrenic Patients
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Rania Hassan Shalby, Lecturer of Oral Medicine, Fayoum University
Other Study IDs: 19038219038211011
Record Dates: First submitted 2023-03-10; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders; Periodontal Diseases
Keywords: schizophrenia; antipsychotics; periodontal disease; hyperprolactinemia
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Periodontal Diseases; Schizophrenia; Hyperprolactinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exposure 1: Schizophrenic patients that have been taking antipsychotic drugs inducing hyperprolactinemia (FGAs and the SGAs; amisulpride, risperidone and paliperidone) for at least 1 year
  Interventions: Drug: antipsychotic drugs inducing hyperprolactinemia
- Exposure 2: Schizophrenic patients that have been taking antipsychotics sparing hyperprolactinemia (In SGAs; clozapine, quetiapine, olanzapine, ziprasidone and aripiprazole) for at least 1 year
- Non exposure (basline): Newly diagnosed schizophrenic patients and/ or patients did not receive any psychiatric treatment for at least 1 year

INTERVENTIONS:
Drug: antipsychotic drugs inducing hyperprolactinemia — not exposed
  Other Names: antipsychotic drugs not inducing hyperprolactinemia
  Groups: Exposure 1

SUMMARY:
The aim of the present cohort retrospective study is to explore the effect of antipsychotics on periodontal health and the possible effect of antipsychotic-induced hyperprolactinemia as a risk factor for periodontal disease progression in schizophrenic patients.

The study population consisted of three groups: Group A (n = 21): schizophrenic patients who have been taking "prolactin inducing" antipsychotics for at least 1 year, Group B (n = 21): schizophrenic patients who have been taking "prolactin sparing" antipsychotics for at least 1 year and Group C (n = 22): newly diagnosed schizophrenic patients and/or patients who did not receive any psychiatric treatment for at least 1 year.

The study groups underwent an assessment of periodontal condition in terms of pocket depth (PD), clinical attachment loss (CAL), gingival recession, tooth mobility, and bleeding on probing (BOP). Also, bone mineral density was evaluated using DEXA scans and the serum prolactin level was measured by automated immunoassay.

DETAILED DESCRIPTION:
Background and objective: The aim of the present cohort retrospective study is to explore the effect of antipsychotics on periodontal health and the possible effect of antipsychotic-induced hyperprolactinemia as a risk factor for periodontal disease progression in schizophrenic patients.

Methods

1. Study design and setting:

   The current study is a cohort retrospective study that will be performed on schizophrenic patients. All subjects will be recruited from the outpatient clinic of the department of Psychiatry-Faculty of Medicine- MUST University. The patients' database from the department of psychiatry will be filtered, and all patients with a diagnosis of schizophrenia according to DSM-IV-TR criteria for schizophrenia and fulfilling eligibility criteria will be contacted. Also, outpatients newly diagnosed with schizophrenia will be included. Those who agree to be enrolled in the study will sign a written informed consent. For patients previously diagnosed with schizophrenia, medication data will be acquired from prescription files, including the type and duration of the prescribed antipsychotic or other medications.

   Psychiatric assessment and recording of demographic variables such as age, gender, duration of psychiatric disease, and type and duration of antipsychotic medication will be performed by the second investigator (EM.A). Then, all subjects will be referred, with their records and files, to the Faculty of Dentistry at ACU University for periodontal assessment and sample collection.
2. Eligibility criteria:

   The included patients are those: 1) with the diagnosis of schizophrenia; 2) over 20 years old; 3) who did not receive any periodontal treatment for the past year; and 4) with at least 20 remaining teeth. To avoid potential confounding factors, the excluded patients are: 1) those with systemic conditions that may affect periodontal status such as; DM, CVS, metabolic syndrome, osteoporosis, AIDS, and chronic alcoholism (3, 4, 17); 2) those with local factors that may aggravate and predispose for periodontal diseases, such as orthodontic and prosthetic appliances, parafunctional habits, and heavy smoking (4, 23-25); and 3) those receiving any systemic medication and/or systemic antibiotics for the past 6 months. Additionally, exclusion criteria involved 4) patients undergoing any type of periodontal treatment for the past year; 5) patients within the childhood and adolescent psychiatry section; and 6) patients who received antipsychotic medication for ≥ 12 months.
3. Estimating the sample size:

   The sample size was calculated considering type I error (α) of 0.05 and power (1-β) of 0.9. Based on a previous study by (16) that used proportions, inequality, and two independent groups (Fisher's exact test) to compare patients with a pocket depth of 4 mm to those with no pocket depth identified in patients receiving antipsychotics 12 months with effect size, the sample size was calculated and found to be a total of 64 patients. The application G*Power 3.1.9.7 [16] was used to determine the sample size needed for the study.
4. Participants:

The study population will be divided into three groups: Exposure groups will be divided according to their "prolactin-inducing" or "prolactin sparing" effect (26-36). Group A (n = 21): schizophrenic patients that have been taking antipsychotic medication that may induce hyperprolactinemia (FGAs and SGAs; amisulpride, risperidone, and paliperidone) for at least 1 year, group B (n = 21): schizophrenic patients who have been taking antipsychotics that do not have a significant effect on serum prolactin levels (in SGAs, clozapine, quetiapine, olanzapine, ziprasidone, and aripiprazole) for at least 1 year and Group C (n = 22): newly diagnosed schizophrenic patients and/or patients who did not receive any psychiatric treatment for at least 1 year.

[4] Outcome measurements: The primary outcome was the assessment of periodontal condition in all study groups measured in terms of pocket depth (PD), tooth mobility, clinical attachment loss (CAL), gingival recession, and bleeding on probing (BOP), while the secondary outcomes were evaluation of BMD and the serum prolactin level (measured by automated immunoassay in ng/ml).

[6]Assessment of clinical data and patient condition: Assessment of mental health: The Positive and Negative Syndrome Scale (PNSS) (37) was used to evaluate each patient's clinical history and current mental health state.

Periodontal evaluation:

All teeth were evaluated and recorded. The means for the following parameters were computed: pocket depth (PD), clinical attachment loss (CAL), and bleeding on probing (BOP) (38, 39). Using a manual periodontal probe (Williams' periodontal probe, PCP-12; Hu-Friedy, Chicago, IL, USA), PD and CAL measurements were collected on six surfaces per tooth (mesio-buccal, mid-buccal, disto-buccal, and mesio-lingual, mid-lingual, disto-lingual, or palatal surface).While CAL measures the distance between the cement-enamel junction of the tooth and the deepest aspect of the pocket, probing pocket depth measures the distance between the gingival margin and the deepest part of the pocket. Total mean PD of the six locations for each tooth was computed for each patient and distance was recorded to the nearest millimeter (40). Sulcus depths between 0 and 2 mm were regarded as normal (41). Gingival recession was measured from the CEJ to the marginal border of the soft tissue on the buccal and lingual sides of each tooth. The total mean number of recessions per tooth for each patient was used to record tooth recessions. Gingival recession, if present, was only used to calculate CAL by its addition to PD.

Four surfaces per tooth were examined for BOP readings (mesial, distal, buccal, and lingual or palatal surface). Bleeding on probing was examined directly after the PD measurement and was reported as absent (0) or present (1). 30 seconds after applying the periodontal probe). The proportion of teeth displaying BOP was recorded.

Generalized mild periodontitis is defined as >30% of remaining teeth with PD 5 mm and 7 mm, as per the 2015 Update to the 1999 Classification of Periodontitis. Severe periodontitis was defined as a probing depth (PD) of 7 mm, with localised periodontitis involving 30% of remaining teeth and generalised periodontitis involving >30% of remaining teeth (42) .

Assessment of bone mineral density:

Dual-energy X-ray absorptiometry (DEXA scan) is an advanced technology that could detect bone mineral density. The GE Lunar Prodigy densitometer was used to perform this test.To determine what constitutes healthy bone, we utilized the World Health Organization's criteria: a T score of -1 indicates normal bone, a T score between -1 and -2.5 indicates osteopaenia, and a T score of -2.5 indicates osteoporosis.

Measurement of serum prolactin level:

Blood will be withdrawn from all patients to determine the fasting serum prolactin level. Prolactin concentrations in blood will be measured in a faculty laboratory by automated immunoassay methodology (43).

7] Data collection and management: Periodontal assessment will be carried out by the primary investigator (S.R.), who will be unaware of the patient's psychological status and records (to avoid potential bias). The third investigator (M.C.) will collect all patient records to perform the final analysis.

STATISTICAL METHODS:

Quantitative (continuous) variables were expressed as mean ± SD. As the quantitative variables were not normally distributed, the Kruskal-Wallis test (a non-parametric test) was used to compare them among the 3 study groups. A post hoc analysis was done for variables that showed a statistically significant difference in the Kruskal-Wallis test using Dwass-Steel-Critchlow-Fligner pairwise comparisons. As for qualitative variables (categorical), the chi-square test was used to compare them among the 3 study groups, and values were expressed as percentages. Also, linear regression analysis was performed to study the relation between 2 quantitative variables (serum prolactin level and PD measurements), while ordinal logistic regression was used to relate one quantitative (serum prolactin level) and one qualitative (BMD or grades of periodontitis) variables.

ELIGIBILITY:
Inclusion Criteria:

1. with the diagnosis of schizophrenia
2. over 20 years old
3. did not receive any periodontal treatment for the past year
4. with at least 20 remaining teeth.

Exclusion Criteria:

1. with systemic condition that may affect periodontal status such as; DM, cardiovascular diseases, metabolic syndrome, osteoporosis, AIDS and chronic alcoholism
2. having local factors that may aggravate and predispose for periodontal diseases such as; orthodontic and prosthetic appliances, parafunctional habits, and heavy smoking
3. receiving any systemic medication and/or systemic antibiotics for the past 6 months.
4. patients undergoing any type of periodontal treatment for the past year and
5. within childhood and adolescence psychiatry section.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: diagnosis of schizophrenia according to DSM-IV-TR criteria for schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Severity of periodontal diseases | 1 months
  The primary outcome will be the assessment of periodontal condition in all study groups measured in terms of Pocket depth (PD), clinical attachment loss (CAL) (both measured using graduated periodontal probe in mm)
gingival condition | 1 months
  bleeding on probing (BOP) using scores from 0-3
tooth mobility | 1 months
  in mm

SECONDARY OUTCOMES:
Serum prolactin level | 1 months
  measurement of serum prolactin level ( measured by automated immunoassay in ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Rania H Shalby, phd, Principal Investigator — Faculty of Dentistry-Fayoum University
Locations (1):
- Rania Hassan Shalby, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No